CLINICAL TRIAL: NCT05399758
Title: Nociception Evaluated by the NOL® Index in Sedated Patients in the Intensive Care Unit
Status: Suspended | Type: Observational
Why Stopped: Technical problems
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Antonello Penna, Principal Investigator, Anesthesiologist, MD-PhD, University of Chile
Other Study IDs: OAIC: 1219/21
Record Dates: First submitted 2022-05-16; First posted 2022-06-01 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Nociceptive Pain; Sedation Complication
Keywords: Nociception; Opioids; Pain monitor
MeSH Terms: conditions — Nociceptive Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU sedated patients: Critical patients sedated with propofol and fentanyl The values obtained with the use of the NOL® index will be recorded and compared with the standard measurements of pain assessment (Behavioral Pain Scale (BPS) and/or CPOT)
  Interventions: Device: NOL monitor

INTERVENTIONS:
Device: NOL monitor — NOL monitor data will be acquired, as well as clinical assessment of pain and fentanyl dosage.

SUMMARY:
Due to their underlying pathology and the necessary complicated procedures to which they are exposed, patients in the intensive care unit experience varying degrees of pain at some point in their evolution. Evidence has established short-term and long-term negative consequences of unresolved pain or excessive analgesic sedation. However, pain assessment or adequate nociceptive monitoring remains a significant challenge, especially in non-communicative patients under deep sedation, who urgently need to expand and improve current tools.

Pain assessment in critically ill patients is challenging; limitations in their ability to communicate (neurocognitive deficit, use of endotracheal tube) or altered consciousness (deep sedation) make them unable to self-report their pain with standard pain scales. The Behavioral Pain Scale (BPS) and the Critical-Care Pain Observation Tool (CPOT) are the pain assessment tools with the best performance and reliability for patients in these conditions.

Different technologies are used to monitor nociceptive responses caused by surgical stress in patients under general anesthesia that together with the clinical evaluation, manage to keep patients in the best analgesic conditions, improving the post-surgical prognosis. In particular, the NOL® nociceptive index (Medasense, Ramat Gan, Israel) is a multiparametric detection of nociception/pain, delivering a dimensionless score (0 -100) calculated through an algorithm (patented) and based on the registry of four biometric sensors (photoplethysmography, galvanic skin response, temperature, and accelerometer). NOL index value between 10-25 is the most appropriate for maintaining analgesia during general anesthesia.

The ease and low invasiveness of this system (all sensors are implemented in a finger clip, similar to an oxygen saturation monitor) may allow its potential use in the context of intensive care unit patients. Some studies have recently been published that highlight the possible usefulness of the NOL® index in critically ill patients. However, in these studies, the assessment of nociception was limited to acute nociceptive procedures only.

DETAILED DESCRIPTION:
In the following protocol, we will study the feasibility of using the NOL® index to evaluate nociception in patients under sedation with propofol and opioid analgesics such as fentanyl.

This study aims to describe the feasibility of using the NOL® nociception index as an objective tool for assessing pain/nociception in patients with sedation in the Intensive Care Unit (ICU).

The values obtained with the use of the NOL® index will be recorded and compared with the standard measurements of pain assessment (Behavioral Pain Scale (BPS) and/or Critical-Care Pain Observation Tool (CPOT)) in patients with a deep/superficial sedation protocol (SAS 1-2). The values obtained after exposure to nociceptive stimuli such as interventions, cleaning, and invasive procedures, among others, will be registered.

In particular, scales such as CPOT and NOL® can be complementary since both measure different components related to pain. The CPOT measures expressive behaviors related to pain, and the NOL measures physiological parameters involved in the process of nociception, which can lead to pain.

Two other aims:

To compare the registration of the NOL® index and the degree of sedation by the BIS® index with variables derived from the processing of the frontal EEG.

To evaluate the effect of sedo-analgesia protocols on the NOL® index. The impact of administering sedation/analgesia protocols with propofol/fentanyl and their effects on the NOL® index will be followed up and evaluated.

ELIGIBILITY:
Inclusion Criteria:

* ICU sedated patients under propofol and fentanyl

Exclusion Criteria:

* Sedation duration less than 72 h
* Stroke
* Opioid user before ICU hospitalization
* Atrial fibrillation
* Pregnancy/lactation
* Patient with antiarrhythmic agents

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients sedated with propofol and fentanyl
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-07-20 (Estimated)

PRIMARY OUTCOMES:
NOL monitor values | Day 3
  Values will be recorded and compared with fentanyl dosage and clinical pain assesment

SECONDARY OUTCOMES:
Fentanyl dosage | Day 3
  Values of fentanyl dosage
Clinical pain assessment (Behavioral Pain Scale) | Day 3
  Values of pain scale
BIS index | Day 3
  Values of BIS index obtained by BIS monitor

CONTACTS AND LOCATIONS:
Locations (2):
- Chile (2):
  - Centro de Investigación Cínica Avanzada (CICA), Hospital Clinico de la Universidad de Chile, Santiago, RM
  - Hospital Clinico de la Universidad de Chile, Santiago, RM

IPD SHARING:
Plan to Share IPD: No